CLINICAL TRIAL: NCT03295747
Title: Peppermint Oil Pharmacokinetics/Dynamics and Novel Biological Signatures in Children With Functional Abdominal Pain
Acronym: PMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Shulman, M.D. (Other)
Responsible Party: Sponsor-Investigator, Robert Shulman, M.D., Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT009101-01 (NIH)
Record Dates: First submitted 2016-12-02; First posted 2017-09-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — peppermint oil

STUDY DESIGN:
Intervention Model Description: Participants randomized to one of three prospective arms as reflected by three treatment doses for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 180 mg (Experimental): 180 mg of peppermint oil
  Interventions: Drug: Peppermint oil
- 360 mg (Experimental): 360 mg of peppermint oil
  Interventions: Drug: Peppermint oil
- 540 mg (Experimental): 540 mg of peppermint oil
  Interventions: Drug: Peppermint oil

INTERVENTIONS:
Drug: Peppermint oil — Three doses of peppermint oil will be investigated: 180, 360, 540 mg; i.e. three arms.
  Other Names: Enteric coated peppermint oil capsules

SUMMARY:
Aim 1 - Determine the pharmacokinetics of PMO (menthol) of three different doses in children with functional abdominal pain (FAP) (n=30).

Aim 2 - Determine pharmacodynamic effect of three different doses of PMO on gut microbiome composition and contractile activity/gut transit rate.

DETAILED DESCRIPTION:
Children with functional abdominal pain (FAP) ages 7-12 years (n=30) will be recruited.

The study participants will be admitted to the Children's Nutrition Research Center. A medical history and a general physical examination performed by the investigator or the research nurse. The height, weight, and vital signs (pulse rate, respiratory rate, and seated blood pressure) will be obtained. After application of a topical anesthetic to the site chosen for study-related blood sampling, a cannula will be inserted e to obtain repeated blood samples.

At approximately 0900, subjects will receive one of three doses of PMO as a single oral dose. Immediately prior to administration of the PMO, a blood sample will be obtained to measure total menthol concentration and leukocytes for isolation of DNA for CYP2A6 and UGT2B7 genotyping.

After PMO administration, repeated blood samples will be obtained over 24 hours.

At 2 hours after PMO administration, participants will be given a standardized meal and will eat ad libitum thereafter.

After completion of the final (24 hours) blood samples, vital signs will be reassessed and the venous cannula removed. Parents will receive a follow-up call from the research coordinator to access/evaluate if any adverse effects from dose or blood sampling received at the overnight study visit.

Prior to and after administration of peppermint oil (PMO) for 1 week at the dose defined above, children will undergo measurement of gut microbiome composition and GI motility and transit time. At the time of the stool collection, the child will also keep a 3 day diet history.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 7-12 years old
2. They will be able to complete the protocol
3. A child will be recruited if the medical evaluation reveals no organic reason for the abdominal pain

Exclusion Criteria:

1. Children who have had past bowel surgery;
2. A child with documented GI disorders (e.g., Crohn's disease);
3. A child with a serious chronic medical condition (e.g., diabetes);
4. A child with a weight and/or height < 2 SD for age;
5. Children with chronic conditions with GI symptoms (e.g., cystic fibrosis);
6. Children with autism spectrum disorder, significant developmental delay, psychosis, depression, or a history of bipolar disorder;
7. Children who have been treated with antibiotics/probiotics within 2 mo. (because of effects on microbiome analysis).
8. Children who speak only Spanish

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 24 hours
  Area under the curve

SECONDARY OUTCOMES:
Contractility | Prior to and during peppermint oil treatment
  Number and amplitude of gut contractions as measured by SmartPill
Gut Microbiome Composition | Prior to and during peppermint oil treatment
  Microbiome is defined for this study as a statistically significant change from baseline after treatment with PMO, correcting for multiple testing (q value). Such changes may occur with respect to gut microbiome diversity and/or composition (e.g., phylum, family, genera). We anticipate there will be an increased bacterial diversity, as well as increases in the abundance of organisms associated with a healthy microbiome, in response to PMO administration.
Motility | Prior to and during peppermint oil treatment
  Gut transit time as measured by SmartPill

CONTACTS AND LOCATIONS:
Overall Officials: Shulman J. Shulman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shulman RJ, Chumpitazi BP, Abdel-Rahman SM, Garg U, Musaad S, Kearns GL. Randomised trial: Peppermint oil (menthol) pharmacokinetics in children and effects on gut motility in children with functional abdominal pain. Br J Clin Pharmacol. 2022 Mar;88(3):1321-1333. doi: 10.1111/bcp.15076. Epub 2021 Oct 19. PMID 34528282
- [Result] Thapa S, Luna RA, Chumpitazi BP, Oezguen N, Abdel-Rahman SM, Garg U, Musaad S, Versalovic J, Kearns GL, Shulman RJ. Peppermint oil effects on the gut microbiome in children with functional abdominal pain. Clin Transl Sci. 2022 Apr;15(4):1036-1049. doi: 10.1111/cts.13224. Epub 2022 Jan 20. PMID 35048535

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03295747/Prot_SAP_000.pdf